CLINICAL TRIAL: NCT04166708
Title: The Footwork Step Technique in Flamenco Dancing: A Case Study
Brief Title: The Footwork Step Technique in Flamenco Dancing
Status: Completed | Type: Observational
Sponsor: Telethusa Centre for Flamenco Research (Other)
Responsible Party: Sponsor
Other Study IDs: 6777
Record Dates: First submitted 2019-11-09; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Kinesics; Kinematics; Injuries
Keywords: Professional Flamenco Dancer; Footwork step; Ground Reaction Force; Center of mass
MeSH Terms: conditions — Kinesics; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A professional flamenco dancer will perform a ZAP 3 test, a sequence of single strikes of the feet performed continuously for 15 sec. Kinetic and kinematic studies will be recorded during the performance.

DETAILED DESCRIPTION:
Flamenco is a highly emotional and sensitive dance, which is one of the most characteristic elements of Spanish culture. It is both physically and mentally demanding, with the emphasis on footwork technical execution and the aesthetic of arms and trunk movements. Years of training are necessary to achieve any level of proficiency as professional flamenco dancer.

Therefore proper execution of the movements minimize the risk of injury accompanying foot - ground contact which was reported by several studies. The most suffering parts of the dancer's body are the cervical and lumbar spine, knee and foot.

Despite the growing number of studies on flamenco dancing, there is a lack of investigations focused on understanding how does the flamenco dancer's body work to mitigate an injury risk. Therefore, the purpose of this study is to examine the parameters related to this issue: vertical Ground Reaction Force, Centre of Mass displacements and knee joint kinematics of the supporting leg They will be registered and analyzed during footwork performance.

A female professional flamenco dancer will perform a footork test called ZAP-3. It is a sequence of single strikes of the feet performed continuously for 15 seconds as fast as possible. 3D lower extremity kinematic data is used to collected using a five-camera motion analysis system (Vicon; Oxford Metrics Ltd., Oxford, UK). Kistler force platform will use to record the Ground reaction forces .

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* More than 15 years as proffesional flamenco dancer.
* More than 20 hours per week dancing flamenco

Exclusion Criteria:

* Not report any musculoskeletal or sub-acute injury prior to 12 months of the study.
* Not report any surgical intervention prior to 12 months of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female profesional flamenco dancer
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Wootwork step test ZAP-3 | 15 seconds
  The participant has to perform ZAP 3 test, a sequence of single strikes of the feet performed continuously for 15 sec.
  The first footwork step is made with the ball of the Foot with the non supporting leg. The second footwork step that will be produced by dropping the heel on the floor and making an audible sound. It is called Heel Drop (HD). The other leg will perform the third footwork step striking only the heel on the floor. The fourth one is made with the other leg, the supporting leg, when the ball of the foot is planted, repeating a HD step footwork. The fifth one is made by the non supporting leg, tapping the tip of the toe on the floor behind the base of support. The last one step is also made with the other leg, the supporting leg, meantime the ball of the foot is planted the heel is dropped on the floor repeating a HD step footwork. Numbers of footwork steps performed will be recorded. A greater number of strokes are associated with a better result.
Centre of mass oscillations | 15 seconds
  During ZAP-3 test, Centre of mass oscillations will be registered. Three-dimensional lower extremity kinematic data are collected using a five-camera motion analysis system at a sampling rate of 120 Hz (Vicon; Oxford Metrics Ltd., Oxford, UK). Body segments were defined according to the Golem model by means of 35 reflective markers attached to the head (4), trunk (4), pelvis (3), arms (7) and legs (5). Centre of mass oscillations will be measured in metres.
Knee joint angular changes | 15 seconds
  During ZAP-3 test, Centre of mass oscillations will be registered. Three-dimensional lower extremity kinematic data are collected using a five-camera motion analysis system at a sampling rate of 120 Hz (Vicon; Oxford Metrics Ltd., Oxford, UK). Body segments were defined according to the Golem model by means of 35 reflective markers attached to the head (4), trunk (4), pelvis (3), arms (7) and legs (5). Knee joint angular changes in the sagittal plane will be registered in degrees.
Ground Reaction Forces | 15 seconds
  The vertical component of Ground Reaction Forces will be measured using Kistler force platform. The subject was asked to perform twice, in order to place both right and left foot on the force platform while performing footwork steps test ZAP-3. Ground Reaction Forces will be registered in degrees in newtons unit.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Vargas-Macías, PhD, Principal Investigator — Telethusa Centre for Flamenco Research
Locations (1):
- Alfonso Vargas-Macías, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Research Projet — http://www.flamencoinvestigacion.es/pi-a1-2015-biomechanics-of-flamenco-dancing/